CLINICAL TRIAL: NCT02497079
Title: Comparison of the Diagnostic Accuracy of Nested and Real-time Polymerase Chain Reaction for Mycobacterium Tuberculosis Using EBUS-TBNA Samples in Patients With Isolated Intrathoracic Lymphadenopathy
Brief Title: Diagnostic Accuracy of Polymerase Chain Reaction for Mycobacterium Tuberculosis Using EBUS-TBNA Samples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Seop Eom, Clinical Assistant Professor, Pusan National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNUH-P-1
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Lymphadenopathy; Tuberculosis; Sarcoidosis
Keywords: Bronchoscopy; Ultrasonography; Tuberculous lymphadenitis; Polymerase chain reaction; Sensitivity and specificity
MeSH Terms: conditions — Lymphadenopathy; Tuberculosis; Sarcoidosis; Tuberculosis, Lymph Node; Hypersensitivity | interventions — Polymerase Chain Reaction; Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nested PCR for formalin-fixed tissues (Experimental): In all patients, nested polymerase chain reaction for Mycobacterium tuberculosis is performed with formalin-fixed paraffin-embedded specimens obtained by endobronchial ultrasound-guided transbronchial needle aspiration.
  Interventions: Device: Nested PCR for formalin-fixed tissues
- Nested PCR for fresh tissues (Experimental): In all patients, nested polymerase chain reaction for Mycobacterium tuberculosis is performed with specimens in sterile saline obtained by endobronchial ultrasound-guided transbronchial needle aspiration.
  Interventions: Device: Nested PCR for fresh tissues
- Real-time PCR for fresh tissues (Experimental): In all patients, real-time polymerase chain reaction for Mycobacterium tuberculosis is performed with specimens in sterile saline obtained by endobronchial ultrasound-guided transbronchial needle aspiration.
  Interventions: Device: Real-time PCR for fresh tissues

INTERVENTIONS:
Device: Nested PCR for formalin-fixed tissues — For nested PCR, formalin-fixed paraffin-embedded tissues were incubated in 1 mL of xylene at 60°C for 30 min and then centrifuged for 10 min. Paraffin and the supernatant were removed from the samples after centrifugation. The same procedures were repeated until deparaffinization was complete. After adding 1 mL of alcohol, the samples were centrifuged for 5 min, and the supernatant was removed. The sample was then air-dried as a pellet. DNA was extracted using QIAamp (Qiagen, Valencia, CA, USA). PCR amplifications were performed using Mycobacterium tuberculosis IS6110 primers. The first round using outer primers and the second round using inner primers amplified a 256- and 181-bp fragment, respectively. Finally, the PCR products were visualized in a 2% agarose gel.
  Other Names: MTB-PCR kit; Biosewoom, Seoul, South Korea
  Arms: Nested PCR for formalin-fixed tissues
Device: Nested PCR for fresh tissues — For nested PCR with specimens in sterile saline, DNA was extracted using QIAamp (Qiagen, Valencia, CA, USA). PCR amplifications were performed using Mycobacterium tuberculosis IS6110 primers. The first round using outer primers and the second round using inner primers amplified a 256- and 181-bp fragment, respectively. Finally, the PCR products were visualized in a 2% agarose gel.
  Other Names: MTB-PCR kit; Biosewoom, Seoul, South Korea
  Arms: Nested PCR for fresh tissues
Device: Real-time PCR for fresh tissues — For real-time PCR, specimens in sterile saline were filtered and 1 mL of phosphate based saline was added. After centrifugation for 3 min, the supernatant was removed. Next, 50 μL of extraction buffer was added to the sample, and the sample was heated at 100°C for 20 min. After centrifugation for 3 min, the supernatant was used in PCR. Real-time PCR was performed using the AdvanSure TB/NTM real-time PCR kit. Three channels were used in the real-time PCR reaction (Mycobacterium tuberculosis complex, mycobacteria, and internal control). Signals for FAM, HEX, and Cy5 were measured in each channel. Mycobacterium tuberculosis was considered present if the cycle threshold of rpoB was less than 35 on each signal and greater than or equivalent to that of IS6110.
  Other Names: AdvanSure TB/NTM real-time PCR kit; LG, Seoul, South Korea
  Arms: Real-time PCR for fresh tissues

SUMMARY:
The purpose of this study is to compare the diagnostic efficacy of nested and realtime polymerase chain reaction for Mycobacterium tuberculosis using EBUS-TBNA samples in patients with isolated intrathoracic lymphadenopathy.

DETAILED DESCRIPTION:
Although endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) has been widely used to perform mediastinal lymph node sampling, little information is available on polymerase chain reaction for Mycobacterium tuberculosis (TB-PCR) using EBUS-TBNA samples in patients with isolated intrathoracic lymphadenopathy. In addition, two methods of TB-PCR (nested PCR and realtime PCR) are available for the detection of Mycobacterium tuberculosis and which method is superior for detection of Mycobacterium tuberculosis has not been established in patients with isolated intrathoracic lymphadenopathy.

Thus, this study was design to compare the diagnostic efficacy of nested and realtime TB-PCR using EBUS-TBNA samples in patients with isolated intrathoracic lymphadenopathy in South Korea, where the incidence of tuberculosis is intermediate (97/100,000 per year).

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated intrathoracic lymphadenopathy

Exclusion Criteria:

* Suspicion of primary lung cancer on CT or PET scan
* Suspicion of pulmonary tuberculosis on CT or PET scan
* Suspicion of sarcoidosis of lung parenchyma on CT or PET scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who detected each polymerase chain reactions for Mycobacterium tuberculosis | 6 months
  In all participants with isolated intrathoracic lymphadenopathy, three modalities of TB-PCR (nested PCR for formalin-fixed paraffin-embedded tissues, nested PCR for fresh tissues and real-time PCR for fresh tissues) are performed using EBUS-TBNA samples. The numbers of participants who reported as positive for each TB-PCR modalities are collected. From these data, sensitivity, specificity and diagnostic accuracy of each TB-PCR modalities to diagnose tuberculous lymphadenitis will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Ha Mok, Master, Principal Investigator — Pusan National University Hospital; Jung Seop Eom, Master, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, Busan, South Korea

REFERENCES:
- [Background] Navani N, Lawrence DR, Kolvekar S, Hayward M, McAsey D, Kocjan G, Falzon M, Capitanio A, Shaw P, Morris S, Omar RZ, Janes SM; REMEDY Trial Investigators. Endobronchial ultrasound-guided transbronchial needle aspiration prevents mediastinoscopies in the diagnosis of isolated mediastinal lymphadenopathy: a prospective trial. Am J Respir Crit Care Med. 2012 Aug 1;186(3):255-60. doi: 10.1164/rccm.201203-0393OC. Epub 2012 May 31. PMID 22652031
- [Background] Navani N, Molyneaux PL, Breen RA, Connell DW, Jepson A, Nankivell M, Brown JM, Morris-Jones S, Ng B, Wickremasinghe M, Lalvani A, Rintoul RC, Santis G, Kon OM, Janes SM. Utility of endobronchial ultrasound-guided transbronchial needle aspiration in patients with tuberculous intrathoracic lymphadenopathy: a multicentre study. Thorax. 2011 Oct;66(10):889-93. doi: 10.1136/thoraxjnl-2011-200063. Epub 2011 Aug 3. PMID 21813622
- [Background] Sun J, Teng J, Yang H, Li Z, Zhang J, Zhao H, Garfield DH, Han B. Endobronchial ultrasound-guided transbronchial needle aspiration in diagnosing intrathoracic tuberculosis. Ann Thorac Surg. 2013 Dec;96(6):2021-7. doi: 10.1016/j.athoracsur.2013.07.005. Epub 2013 Sep 12. PMID 24035300
- [Background] Statement on sarcoidosis. Joint Statement of the American Thoracic Society (ATS), the European Respiratory Society (ERS) and the World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) adopted by the ATS Board of Directors and by the ERS Executive Committee, February 1999. Am J Respir Crit Care Med. 1999 Aug;160(2):736-55. doi: 10.1164/ajrccm.160.2.ats4-99. No abstract available. PMID 10430755
- [Background] Bezabih M, Mariam DW, Selassie SG. Fine needle aspiration cytology of suspected tuberculous lymphadenitis. Cytopathology. 2002 Oct;13(5):284-90. doi: 10.1046/j.1365-2303.2002.00418.x. PMID 12421444